CLINICAL TRIAL: NCT06102668
Title: Long-term Survival and Parenteral Nutrition Dependence in Adult Patients With Non-malignant Short Bowel Syndrome
Brief Title: Survival and PN Dependence in SBS Patients
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Collaborators: Jinling Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: FirstAHUSTChina
Record Dates: First submitted 2023-10-21; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Short bowel syndrome (SBS) is a rare condition resulting from the loss of portions of the small intestine, and can cause a spectrum of metabolic and physiologic disturbances.The objective of this study was to determine the longterm survival and parenteral nutrition dependence of adult patients with SBS.

DETAILED DESCRIPTION:
Short bowel syndrome (SBS), the most common form of intestinal failure, is a rare condition resulting from the loss of portions of the intestine, typically because of extensive surgical resection or loss of intestinal function. Patients with SBS often stuffer from intestinal insufficiency or intestinal failure because they are unable to maintain fluid and nutrient balances on a normal diet. SBS can cause various metabolic and physiologic disturbances. Although parenteral nutrition is a life-saving measure for many patients with SBS, patients with SBS is associated with decreased survival and parenteral nutrition (PN) dependence. Few studies have reported the survival and PN dependence in adult SBS patients in China.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with SBS.

Exclusion Criteria:

* age <18 years; patients with active malignant tumors.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SBS caused by extensive bowel resection with a remnant small intestine length of <200cm.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Survival | 2012/1/1-2019/1/1
  Survival rate in patients with SBS
Parenteral nutrition dependence | 2012/1/1-2019/1/1
  Parenteral nutrition dependence in patients with SBS

SECONDARY OUTCOMES:
Risk factors | 2012/1/1-2019/1/1
  Risk factors of mortality and parenteral dependence in patients with SBS
Cause of death | 2012/1/1-2019/1/1
  Cause of death in patients with SBS at the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: JIANFENG GONG, M.D., Principal Investigator — Jinling Hospital, China

IPD SHARING:
Plan to Share IPD: Undecided